CLINICAL TRIAL: NCT05158569
Title: Effectiveness of Diaphragmatic Breathing vs. Slow Breathing Techniques on Blood Pressure and Health-related Quality of Life in Adults With Stage 1 Hypertension
Brief Title: Comparison of Breathing Exercise for Hypertensive Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rec/01091 Kamran khan
Record Dates: First submitted 2021-12-13; First posted 2021-12-15 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Hypertension
Keywords: Stage 1 hypertension; Diaphragmatic breathing; Slow breathing; Quality of life
MeSH Terms: conditions — Hypertension; Hypoventilation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Slow breathing exercise group (Experimental): Slow breathing 5-6 breaths/minute, 3 sets of 5 minutes 2 times/day for 4 weeks.
  Interventions: Other: Slow breathing exercise group
- Diaphragmatic breathing exercise group (Experimental): Diaphragmatic breathing, 3 sets of 5 minutes 2 times/day for 4 weeks.
  Interventions: Other: Diaphragmatic breathing exercise group

INTERVENTIONS:
Other: Slow breathing exercise group — The patient will be first asked to close one nostril with a thumb and slowly breathe in completely through the other for 6 seconds. This nostril will be then closed and the patient will exhale through the other nostril over a period of 6 seconds. These steps complete one breathing cycle. An attempt will be made to keep the breathing rate is about 5-6 breaths per minute. Such alternate nostril breathing cycles will be repeated continuously for a period of about 15 minutes (3 sets of 5 minutes) in one sitting.
  Arms: Slow breathing exercise group
Other: Diaphragmatic breathing exercise group — Patients would be instructed to Sit or lie down in a comfortable place and put their hands on their belly.
  Relax the muscles in their neck and shoulders. Breathe in slowly through the nose, keeping their mouth closed. Feel the lungs fill with air and inflate like a balloon while their belly moves outward. Such breathing cycles will be repeated continuously for a period of about 15 (3 sets of 5 minutes) minutes in one sitting.
  Arms: Diaphragmatic breathing exercise group

SUMMARY:
To determine the Effectiveness of diaphragmatic breathing vs. slow breathing techniques on blood pressure and Quality of life in adults with stage 1 hypertension. In accessible literature limited data was found on the comparison of different breathing techniques. The current study will compare the effect of slow vs. diaphragmatic breathing exercises and will demonstrate which one is more effective.

DETAILED DESCRIPTION:
Literature reports that inspiratory muscle training is more effective in reducing Blood Pressure and voluntary diaphragmatic breathing at 10 or 6 breaths per minute for 10 min twice a day for 4 weeks is effective in producing positive outcomes in hypertensive patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient having stage 1 hypertension, Diagnosed after 1 week BP charting

Exclusion Criteria:

* Patients taking antihypertensive medication Patient having comorbidities Smokers and women taking oral contraceptives

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | 4 weeks
  Blood pressure is measured in millimeters of mercury (mm Hg). A blood pressure measurement has two numbers: The top number (systolic) is the pressure of the blood flow when your heart muscle contracts, pumping blood. The bottom number (diastolic) is the pressure measured between heartbeats. The patients are classified according to the range as follows. Hypertension stage 1 SYSTOLIC (mm of Hg): 121-139 DIASTOLIC (mm of Hg): 81-89

SECONDARY OUTCOMES:
Health related Quality of life | 4 weeks
  Measured through EuroQOL-five-dimensional-three-level (EQ-5D-3L) questionnaire which comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems.

CONTACTS AND LOCATIONS:
Overall Officials: Mehwish Waseem, MSPT(CPPT), Principal Investigator — Riphah International University
Locations (1):
- Zakir khan shaheed hospital matta, Swāt, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jones CU, Sangthong B, Pachirat O, Jones DA. Slow breathing training reduces resting blood pressure and the pressure responses to exercise. Physiol Res. 2015;64(5):673-82. doi: 10.33549/physiolres.932950. Epub 2015 Mar 24. PMID 25804100
- [Background] Janet SK, Mangala Gowri P. Effectiveness of deep breathing exercise on blood pressure among patients with hypertension. Int J Pharma Bio Sci 2017; 8(1):B256-60.
- [Background] Ma X, Yue ZQ, Gong ZQ, Zhang H, Duan NY, Shi YT, Wei GX, Li YF. The Effect of Diaphragmatic Breathing on Attention, Negative Affect and Stress in Healthy Adults. Front Psychol. 2017 Jun 6;8:874. doi: 10.3389/fpsyg.2017.00874. eCollection 2017. PMID 28626434